CLINICAL TRIAL: NCT04198987
Title: Dietary Monosaccharide Supplementation in Patients With Congenital Disorders of Glycosylation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David R. Deyle, Principal Investigator, Mayo Clinic
Other Study IDs: 18-007276
Record Dates: First submitted 2019-12-08; First posted 2019-12-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-01

CONDITIONS: Congenital Disorder of Glycosylation
MeSH Terms: conditions — Congenital Disorders of Glycosylation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Researchers are trying to assess whether the use of simple sugars given as a daily dietary supplement can improve the health of children with congenital disorders of glycosylation (CDG).

DETAILED DESCRIPTION:
The goal of this study is to collect data from patients diagnosed with congenital disorders of glycosylation and taking a simple sugar supplement. The study team wants to expand the evidence on the beneficial effects of this treatment in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a biochemically and genetically proven congenital disorder of glycosylation
* Patient is receiving (or planning to receive) oral simple sugar supplementation

Exclusion Criteria:

* Aldolase B deficiency
* Galactosemia
* Hemolytic uremic syndrome
* Severe anemia
* Galactose intolerance

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: We will enroll patients diagnosed with congenital disorders of glycosylation and started on oral simple sugar supplements as part of their routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Measuring effects of oral monosaccharide supplements through growth measurements | length of study, up to 2 years
  To assess the effects of oral monosaccharide supplementation for each participant, changes in participant growth parameters, as well as blood sugar levels, coagulation parameters, liver function, and other measures of organ system function (as appropriate for the specific type of CDG) will be correlated with biomarkers derived from participant blood and urine samples obtained at key time points and then compared to standard normative ranges of data for each measure.
Measuring effects of oral monosaccharide supplements through blood sugar levels | length of study, up to 2 years
  To assess the effects of oral monosaccharide supplementation for each participant, changes in participant growth parameters, as well as blood sugar levels, coagulation parameters, liver function, and other measures of organ system function (as appropriate for the specific type of CDG) will be correlated with biomarkers derived from participant blood and urine samples obtained at key time points and then compared to standard normative ranges of data for each measure.
Measuring effects of oral monosaccharide supplements through liver function results | length of study, up to 2 years
  To assess the effects of oral monosaccharide supplementation for each participant, changes in participant growth parameters, as well as blood sugar levels, coagulation parameters, liver function, and other measures of organ system function (as appropriate for the specific type of CDG) will be correlated with biomarkers derived from participant blood and urine samples obtained at key time points and then compared to standard normative ranges of data for each measure.
Measuring effects of oral monosaccharide supplements through coagulation results | length of study, up to 2 years
  To assess the effects of oral monosaccharide supplementation for each participant, changes in participant growth parameters, as well as blood sugar levels, coagulation parameters, liver function, and other measures of organ system function (as appropriate for the specific type of CDG) will be correlated with biomarkers derived from participant blood and urine samples obtained at key time points and then compared to standard normative ranges of data for each measure.

CONTACTS AND LOCATIONS:
Overall Officials: David Deyle, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to PI's decision.
Supporting Information: Study Protocol
Time Frame: length of study

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials